CLINICAL TRIAL: NCT01073839
Title: Adjuvant Treatment of Resectable Cholangiocellular Carcinoma (CCC) With Cisplatin Plus Gemcitabine. A Prospective Single Center Phase Ib-II Study.
Brief Title: Adjuvant Cisplatin Plus Gemcitabine in Operable Cholangiocellular Carcinoma.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Bernhard Pestalozzi, Prof. Dr. med., University of Zurich
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONK USZ 001-2008
Record Dates: First submitted 2009-06-25; First posted 2010-02-23 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Cholangiocellular Carcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cisplatin plus Gemcitabine (Experimental): Patients after resection of cholangiocellular carcinoma will be allocated to treatment with cisplatin plus gemcitabine.
  Interventions: Drug: Cisplatin and Gemcitabine

INTERVENTIONS:
Drug: Cisplatin and Gemcitabine — Cisplatin 25 mg/m2 days 1 and 8; next cycle starting day 22. Gemcitabine 1000 mg/m2 days 1 and 8; next cycle starting day 22. Total of 8 cycles.
  Other Names: Gemzar; Platinol

SUMMARY:
OBJECTIVES

Primary objective:

The primary objective of the trial is to determine the safety of adjuvant treatment with cisplatin plus gemcitabine for a period of 6 months after curative resection of cholangiocellular carcinoma

Secondary objectives:

Secondary objectives of the trial are to assess the feasibility and efficacy of the adjuvant therapy and to determine duration of response and patterns of failure compared to historical controls without postoperative treatment

Exploratory objectives:

To obtain blood samples and tumor tissue after resection for establishment and characterization of new cholangiocarcinoma cell lines and tumor antigens. Other aims are identification of tumor specific antibodies from blood samples, and characterization of tumor antigens with consecutive development of new specific immunological therapies, e.g. cancer-testis antigens (CTA) for tumor vaccination.

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria

1. Histologically or cytologically confirmed adenocarcinoma of biliary tract (intrahepatic and hilar tumors). Carcinomas involving the gall bladder are allowed.
2. Macroscopically complete resection within 8 weeks before start of chemotherapy.
3. Written informed consent.
4. Health status: WHO performance status (PS) 0-1
5. Age >18 years
6. Adequate renal function (creatinine clearance ≥ 60 ml/min, calculated according to the formula of Cockcroft-Gault)
7. Adequate hepatic function (bilirubin ≤ 3 x LUN, AP ≤ 5 x LUN, ASAT ≤ 5 x LUN)
8. Adequate hematologic function: neutrophils ≥ 1.5 x 109/l, platelets ≥ 100 x 109/l, Hb ≥ 9,5 mg/dl
9. Patient compliance and geographic proximity allowing proper staging, treatment and follow-up.
10. Women who are not breastfeeding and are using effective contraception if sexually active, who are not pregnant and agree not to become pregnant during participation in the trial or during the 12 months thereafter. A negative pregnancy test before inclusion into the trial is required for women < 50 years. Men who agree not to father a child during participation in the trial or during the 12 months thereafter.

Exclusion criteria

1. Pregnancy or breastfeeding women
2. Previous malignancy within 5 years or concomitant malignancy, except: non-melanomatous skin cancer or adequately treated in situ cervical cancer
3. neutrophils < 1.5 x 109/l, platelets < 100 x 109/l, Hb < 9,5 mg/dl
4. bilirubin > 3 x LUN, ALAT > 5 x LUN, ASAT > 5 x LUN
5. Creatinine clearance < 60 ml/min, calculated according to the formula of Cockcroft-Gault
6. Prior chemotherapy with gemcitabine
7. Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV, unstable angina pectoris, history of myocardial infarction in the last 3 months, significant arrhythmias)
8. Psychiatric disorder precluding understanding of information of trial related topics and giving informed consent
9. Active uncontrolled infection
10. Preexisting peripheral neuropathy (> grade 1)
11. Serious underlying medical condition (judged by the investigator) which could impair the ability of the patient to participate in the trial (e.g. uncontrolled diabetes mellitus, active autoimmune disease)
12. Concurrent treatment with other experimental drugs or other anti-cancer therapy; treatment in a clinical trial within 30 days prior to trial entry
13. Known hypersensitivity to the study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Occurence of Grade 3 or 4 toxicities according to NCI-common terminology criteria for adverse events v3.0 | One year

SECONDARY OUTCOMES:
Disease-free survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland

REFERENCES:
- [Derived] Siebenhuner AR, Seifert H, Bachmann H, Seifert B, Winder T, Feilchenfeldt J, Breitenstein S, Clavien PA, Stupp R, Knuth A, Pestalozzi B, Samaras P. Adjuvant treatment of resectable biliary tract cancer with cisplatin plus gemcitabine: A prospective single center phase II study. BMC Cancer. 2018 Jan 11;18(1):72. doi: 10.1186/s12885-017-3967-0. PMID 29325521